CLINICAL TRIAL: NCT06694571
Title: STARS (Sun Protection and Tanning Awareness in Rural Schools)
Brief Title: Sun Protection and Tanning Awareness in Rural Schools
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Tammy Stump, Visiting Instructor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 174239
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2024-10

CONDITIONS: Melanoma; Adolescents
Keywords: prevention; school-based intervention; skin cancer; adolescents; rural health
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Skin cancer prevention education (Experimental): Program components of a rural-adapted skin cancer prevention intervention (i.e., education, action planning exercise, risk assessment activity) will be co-implemented by the research team and participating school staff during a single- or double-session, in-class visit lasting up to 90 minutes. Students will be asked to complete surveys at baseline and one month post-intervention.
  Interventions: Behavioral: Skin cancer prevention educational presentation and activities

INTERVENTIONS:
Behavioral: Skin cancer prevention educational presentation and activities — An intervention visit, lasting up to 90 minutes, will take place during fall, immediately following completion of a baseline survey. This intervention visit may be divided into 2 days, depending on the length of the class periods at the participating schools. During the intervention visit, participants will receive general education on skin cancer and skin cancer prevention, complete a skin cancer risk self-assessment tool, and create a sun protection action plan for an outdoor activity.
  One month later, participants will receive a brief (15-minute) post-intervention survey via email and/or text.

SUMMARY:
Drawing from prior school-based skin cancer prevention programs, we have adapted intervention materials to target rural high schoolers. Program components (including in-class education) will be co-implemented by the research team and participating school staff, with a focus on sustainability beyond the immediate study period. Interviews and surveys following initial implementation will evaluate both the effectiveness of the program.

DETAILED DESCRIPTION:
The STARS study pilot tests a skin cancer prevention intervention adapted for use in rural schools. Participants will be recruited from approximately 14 districts in Utah. We have established collaborations with schools, districts, and the Utah State Board of Education (USBE) and they are committed to partnering with us on this project.

The research coordinator will contact district-level officials who will be asked to express their support of the study when facilitating the coordinator's contact with school principals and teachers (e.g., health teachers, science teachers). The research coordinator will also directly contact school principals and teachers to discuss participation in the study.

An intervention visit, lasting up to 90 minutes, will take place immediately following completion of a baseline survey. This intervention visit may be divided into 2 days, depending on the length of the class periods at the participating schools. During the intervention visit, students will receive general education on skin cancer and skin cancer prevention, complete a skin cancer risk self-assessment tool, and create a sun protection action plan for an outdoor activity.

One month later, participants will receive a brief (15-minute) post-intervention survey via email and/or text.

ELIGIBILITY:
Inclusion Criteria:

* Students are eligible if they are enrolled in a Utah high school (e.g. grades 9-12).

Exclusion Criteria:

* None

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Sun protection index scores | Baseline, One month
  Surveys (a baseline and a 1 month follow-up) will be distributed to students to assess changes in sun protection and tanning behaviors as well as knowledge and attitudes about skin cancer prevention. The outcome variable is the students' responses on these surveys and how their responses change over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share deidentified self-report responses to surveys.
Supporting Information: ICF
Time Frame: 4/1/2025-4/1/2028
Access Criteria: These data will be available upon request to the principal investigator, Tammy Stump, Tammy.stump.hci.utah.edu. Data will be shared with other investigators who propose specific aims/hypotheses in order to identify the data elements required.